CLINICAL TRIAL: NCT05552339
Title: SMART-Finder - Identification of Patients With Elevated UACR Levels in a T2DM Cohort
Brief Title: A Study Called SMART-Finder to Look for People With Increased Amounts of Albumin in the Urine (UACR Level) in a Group of Type 2 Diabetes Mellitus Patients
Acronym: SMART-Finder
Status: Recruiting | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 22280
Record Dates: First submitted 2022-09-21; First posted 2022-09-23 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Type 2 Diabetes Mellitus; Chronic Kidney Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic | interventions — finerenone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Type 2 Diabetes Mellitus patients: MyTherapy App users with Self-reported Type 2 Diabetes Mellitus who had been prescribed drugs for their T2DM.
  Interventions: Drug: Finerenone (Kerendia, BAY94-8862); Drug: Type 2 DM drugs

INTERVENTIONS:
Drug: Finerenone (Kerendia, BAY94-8862) — Following the physicians' decision.
Drug: Type 2 DM drugs — Following the physicians' decision

SUMMARY:
This is an observational study in which data from people with type 2 diabetes mellitus (T2DM) in Germany who use the medical app "myTherapy" are studied.

In observational studies, only observations are made without specified advice or interventions.

In people with T2DM, the body does not make enough of a hormone called insulin or does not use insulin well enough. The resulting high blood sugar level can cause damage to the kidneys over time. As a result, chronic kidney disease (CKD) can occur as a complication of T2DM.

Kidneys filter extra water and waste out of the blood and make urine. CKD is a long-term, progressive decrease in the kidneys' ability to properly filter the blood. Abnormal amounts of proteins such as albumin in the urine are a sign of kidney damage, as proteins are normally kept in the blood.

The amount of albumin in the urine is measured as so-called urine-albumin-creatinine-ratio (UACR) in this study.

Studies in people with T2DM and CKD in a real-world care setting are limited, particularly those that look at the number of people concerned over time.

The main purpose of this study is to learn how many people with T2DM have also increased amounts of albumin in the urine (UACR level) in users of the medical app "myTherapy" in Germany. In addition, researchers want to learn how these albumin levels change over time.

To answer this, the researchers will collect the participant's UACR level at start of the study and about 12 months later. The UACR is measured by the participant's physician during routine care using urine dip-sticks.

All participants of this study are already receiving or will receive one of the available T2DM treatments prescribed by their doctors according to the approved use or are regularly using devices to check their blood sugar levels. And they use the "myTherapy" app to support and track their T2DM therapy.

The data collected includes both participant-reported data and physician-provided lab values. All data are entered into the "myTherapy" app by the participant. They will be collected from October 2022 to December 2024 and cover a period of up to 15 months per participant. Besides this data collection, no further tests or examinations are planned in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients participating in the Chronic Kidney Disease (CKD) awareness program within myTherapy App
* Patient self-reported diagnosis of Type 2 Diabetes Mellitus
* Patients tracking their adherence for at least one of the following drug containing medical products/devices within myTherapy App: Metformin, Acarbose, Dipeptidyl peptidase (DDP)-4 inhibitors, Glucagon-like peptide (GLP) inhibitors, RAS inhibitors, Sodium-dependent glucose transporters 2 (SGLT2) inhibitors, Basal insulin, Finerenone (once available in Germany), Sulfonylurea, Glucose test strips
* Adult (≥ 18 years) female, male or diverse patient
* Signed informed consent

Exclusion Criteria:

* Patient self-reported diagnosis of Type 1 Diabetes Mellitus
* Patients tracking their adherence for at least one of the following medical products: Insulin pump

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MyTherapy App users in Germany with the Self-reported Type 2 Diabetes Mellitus patients who have been prescribed the drugs defined according inclusion criteria will be eligible to be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2023-08-18 (Actual); Primary Completion 2025-11-18 (Estimated); Study Completion 2025-11-18 (Estimated)

PRIMARY OUTCOMES:
Number of patients with Urine albumin-creatinine ratio (UACR) values between 30 and 299 mg/g and above 300 mg/g | Up to 15 months after the date the initial UACR test took place
  The urine albumin-creatinine ratio (UACR) measured by a healthcare professional and provided to the patient

SECONDARY OUTCOMES:
Number of patients changing their UACR values regarding their baseline Albumin-Creatinine-Ratio (ACR) classification. | Up to 15 months after the date the initial UACR test took place
Number of patients with hypertension and nephrotoxic co-medication | 12 month previous informed consent date until end of observation
Mean EuroQol-5 Dimensions (EQ-5D) | Up to 15 months after the date the initial UACR test took place
Diabetes Treatment Satisfaction Questionnaire (DTSQ) | Up to 15 months after the date the initial UACR test took place
Number of patients with CKD, Hypertension, Type 2 Diabetes Mellitus and tobacco use | Up to 15 months after the date the initial UACR test took place
Adherence - number of patients compliant and persistent in the observation period | 12 month previous informed consent date until end of observation
  Patients included:
  1. documenting at least 80% of the expected medication tracked in myTherapy App (compliance), and
  2. not stopping using their medication (persistence).
Number of Health Care Professionals (HCPs) providing UACR to patients | Up to 15 months after the date the initial UACR test took place
Location of HCP | Up to 15 months after the date the initial UACR test took place

CONTACTS AND LOCATIONS:
Locations (1):
- Many locations, Multiple Locations, Germany

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.